CLINICAL TRIAL: NCT02496169
Title: A Prospective, Multi-centric, Nonrandomised Interventional Study of a Sirolimus-eluting Stent With a Biodegradable Polymer for Percutaneous Coronary Revascularization
Brief Title: Prospective multicEntric NonranDomized Registry
Acronym: ExPEND
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eucatech AG (Industry)
Collaborators: CERES GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: eucaLimus2015
Record Dates: First submitted 2015-07-02; First posted 2015-07-14 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Coronary Artery Disease
Keywords: PTCA; stenosis; sirolimus; stent
MeSH Terms: conditions — Coronary Artery Disease; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- eucaLimus (Experimental): Percutaneous Coronary Intervention (PCI)
  Interventions: Device: eucaLimus

INTERVENTIONS:
Device: eucaLimus — Percutaneous Coronary Intervention (PCI)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the eucaLimus Sirolimus Eluting stent system in patients with de novo coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥18 years or the minimum age required for legal adult consent in the country of enrollment.
2. Subject is an acceptable candidate for Percutaneous Coronary Intervention (PCI).
3. Subject is an acceptable candidate for Emergent Coronary Artery Bypass Grafting (CABG).
4. Subject has clinical evidence of ischemic heart disease, stable or unstable angina pectoris or documented silent ischemia.
5. Subject is eligible for dual anti-platelet therapy treatment with aspirin plus either clopidogrel, prasugrel, ticagrelor or ticlopidine.
6. Subject has provided written informed consent.
7. Subject is willing to comply with study follow-up requirements.

Each target lesion/vessel must meet all of the following angiographic criteria for the subject to be eligible for the trial:

1. Subject has up to 3 target lesions in up to 3 separate target vessels Subject has up to 3 target lesions in in up 2 separate target vessels (2 target lesions in 1 vessel and 1 target lesion in a separate vessel). Subject has 1 target lesions in 1 vessel.
2. Target lesion must be de novo.
3. Target lesion must be in major coronary artery or branch (target vessel).
4. Target lesion must have angiographic evidence of ≥ 50% and < 100% stenosis (by operator visual estimate)
5. Target lesion must be ≤ 35 mm in length by operator visual estimate.
6. Target vessel Reference Vessel Diameter (RVD) of 2.25mm - 4.00mm by operator visual estimate.
7. Target lesion must be treatable with a maximum of 1 stents

Exclusion Criteria:

1. Subject has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute ST elevation myocardial infarction (STEMI) within 72 hours prior to the index procedure. Hemodynamically stable non-STEMI (NSTEMI) subjects are eligible for study enrollment.
2. Subject is presenting cardiogenic shock.
3. Subject is pregnant and/or breastfeeding or intends to become pregnant during the duration of the study.
4. Subject has a known allergy to contrast medium that cannot be adequately pre-medicated, or any known allergy to thienopyridine, aspirin, both heparin and bivalirudin, L-605 cobalt-chromium (Co-Cr) alloy or one of its major elements (cobalt, chromium, tungsten and nickel), Polylactic-Co-Glycolic Acid (PLGA), sirolimus
5. Revascularization of any target vessel within 9 months prior to the index procedure or previous PCI of any non-target vessel within 30 days prior to the index procedure.
6. Planned treatment of a lesion not meeting angiographic inclusion and exclusion criteria during the index procedure or after the index procedure.
7. Planned surgery within 6 months of index procedure unless dual antiplatelet therapy can be maintained throughout the peri-surgical period.
8. History of a stroke or transient ischemic attack (TIA) within 6 months prior to the index procedure.
9. Subjects with active bleeding disorders, active coagulopathy, or any other reason, who are ineligible for Dual Antiplatelet Therapy (DAPT).
10. Subject will refuse blood transfusions.
11. Subject has documented left ventricular ejection fraction (LVEF) < 30% within 90 days prior to the index procedure.
12. Subject is dialysis-dependent.
13. Subject has impaired renal function (i.e., blood creatinine > 2.5 mg/dL or 221 μmol/L determined within 7 days prior to the index procedure).
14. Subject has leukopenia (i.e. < 3,000 white blood cells/mm3), thrombocytopenia (i.e. < 100,000 platelets/mm3) or thrombocytosis (i.e. > 700,000 platelet/mm3).
15. Subject is receiving oral or intravenous immunosuppressive therapy (inhaled steroids are permitted), or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus; diabetes mellitus is permitted).
16. Subject is receiving chronic anticoagulation (e.g. coumadin, dabigatran, apixaban, rivaroxaban or any other agent).
17. Subject has life expectancy of < 1 year.
18. Subject is participating in another investigational (medical device or drug) clinical study. Subjects may be concurrently enrolled in a study, as long as the study device, drug or protocol does not interfere with the investigational treatment or protocol of this study.
19. In the investigator's opinion, subject will not be able to comply with the follow-up requirements.

Subjects will be excluded from the trial if any of the target lesions/vessels meets any of the following angiographic criteria:

1. Target lesion is located within a saphenous vein graft or arterial graft.
2. Target lesion involves a side branch of > 2.0 mm in diameter. Note: Lesions within 3 mm of the origin of the right coronary artery may be treated.
3. Target vessel/lesion is excessively tortuous / angulated or is severely calcified, that would prevent complete inflation of an angioplasty balloon. This assessment should be based on visual estimation.
4. Target vessel has angiographic evidence of thrombus.
5. Target vessel was treated with brachytherapy any time prior to the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Target Lumen Revascularisation (TLR) | 12 months post procedure
  Clinical driven TLR

SECONDARY OUTCOMES:
Target Lumen Revascularisation (TLR) | 1 month, 6 months, 24 months post procedure
  Clinical driven TLR
Composite of cardiac death | 1 month, 6 months, 12 months, 24 months post procedure
  MI attributed to the target vessel and clinically driven target lesion revascularization
Composite of all-cause mortality | 24 months post procedure
  any MI and any revascularization, target vessel revascularization or revascularization of nontarget vessels
Stent thrombosis | 1 month, 6 months, 12 months, 24 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Pernes, Dr., Principal Investigator — Hôpital privé d' Antony 1 rue Velpeau 92160 Antony, France